CLINICAL TRIAL: NCT03617926
Title: A Randomized, Controlled, Investigator-Assessor Blinded, Comparative Study to Evaluate the Safety and Efficacy of a Water-Soluble Head Lice Suffocation Product (X92001666) vs RID Shampoo (Pyrethrin) in Subjects With Head Lice
Brief Title: A Clinical Trial to Evaluate Efficacy and Safety of a Water-soluble Head Lice Product.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OYS007-0017
Record Dates: First submitted 2018-07-23; First posted 2018-08-07 (Actual); Results first posted 2022-06-07 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Head Lice; Pediculosis Capitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Test product (Experimental): Water-based lotion (internal code (X92001666)
  Interventions: Device: X92001666
- Reference (Active Comparator): Commercial, pyrethrin-based shampoo (RID shampoo)
  Interventions: Other: RID shampoo

INTERVENTIONS:
Device: X92001666 — the X92001666 product is a lotion to be applied on dry hair for 15 minutes and then washed out using shampoo. The product is to be applied on Day 0 and repeated again on Day 7.
  Other Names: Test product
  Arms: Test product
Other: RID shampoo — Active Comparator: RID shampoo The RID shampoo is to be applied on dry the hair for 10 minutes and then rinsed out with water. the product is to be applied on Day 0 and repeated again on Day 7.
  Other Names: Reference
  Arms: Reference

SUMMARY:
The present study is set-up to compare in vivo clinical performance and safety of the test product versus an in the US commercially available, pyrethrum-based product (RID® shampoo).

DETAILED DESCRIPTION:
The present study is set-up to compare in vivo clinical performance and safety of the test product versus an in the US commercially available, pyrethrum-based product (RID® shampoo). The study will be performed in subjects ≥2 year of both genders with confirmed diagnosis of head lice infestation. To support safety, local and global tolerability, skin and ocular irritation will be assessed and adverse events (AEs) will be registered.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: male / female.
2. Women of childbearing potential is a premenopausal female that is anatomically and physiologically capable of becoming pregnant following menarche.

   Female subjects: are women of childbearing potential who test negative for pregnancy and agree to use a reliable method of birth control or remain abstinent during the study. Methods of contraception considered acceptable include oral contraceptives, contraceptive patch, intrauterine device, vaginal ring, diaphragm with contraceptive gel, or condom with contraceptive gel
   * or are women of non-childbearing potential, defined as: women who have had surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation),
   * or women who are ≥60 years of age.
3. Age: ≥ 2 year of age at the time of enrollment.
4. Subject must have an active head lice infestation defined as at least 5 live lice (adults and/or nymphs) and 5 apparently live nits, present on the scalp and/or hair, as determined by a trained evaluator.
5. Subject is in good general health based on medical history.
6. The subject or his/her parent/legal guardian must give written informed consent, after having been oral and written informed about benefits and potential risks of the trial, as well as information regarding the insurance, taken out to cover the subjects participating in the study. A caregiver must sign an informed consent agreement for children not old enough to do so. Children ages 6-18 years of age will be administered a child's assent form. Subject or his/her parent/legal guardian must be capable of understanding and providing written informed consent.
7. Following application and rinsing of the test products, subject agrees not to shampoo, wash, or rinse their hair or scalp until the 24-hour post treatment evaluation has been completed.
8. The subject agrees not to cut or chemically treat their hair while participating in the study.
9. No more than one working male per household may be excluded from evaluation if he is assessed as being lice free by himself or caregiver.
10. Subject agrees to follow all study instructions, including attending all follow-up appointments.
11. Agree to not use any other pediculicides or medicated hair grooming products for the duration of the study (through Day 10 visit).
12. The parent or legal guardian of a child must be willing to have other family members screened for head lice. If other household members are found to have head lice and are eligible, they must be either enrolled in the study OR receive the standard of care at the site and in the same manner as study participants.
13. Have a single place of residence.
14. The subject or his/her parent or legal guardian must give written informed consent, after having been oral and written informed about benefits and potential risks of the trial, as well as details of the insurance taken out to cover the subjects participating in the study
15. Subjects must agree to not use any other ant-lice treatment for the duration of the study

Exclusion Criteria:

1. Application of any form of head lice treatment, whether prescription or over-the-counter (OTC), or home remedy for 30 days prior to their screening visit (Day 1).
2. Application of any topical medication of any kind on the hair for a period of 48 hours prior to the screening visit.
3. Use of systemic or topical drugs or medications, including systemic antibiotics, which in the opinion of the investigative personnel may interfere with the study results.
4. Known skin allergies, multiple drug allergies or multiple allergies to cosmetic products.
5. History of allergy or hypersensitivity to ragweed, active ingredients or constituents of the test products.
6. Subject with any visible skin/scalp condition at the treatment site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test product.
7. Subjects with chronic scalp disorder.
8. Subject or his/her legal guardian who, in the opinion of the investigative personnel, do not understand the subject requirements for study participations and/or may be likely to exhibit poor compliance with the required visits.
9. Females who are pregnant or nursing.
10. Hair longer than mid-back.
11. Subject suspected or known not to follow instructions
12. Previous participation in this study or participation in any other investigational trial within the preceding 30 days
13. The subject is directly affiliated to the investigator site personnel and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
14. The subject is an Oystershell employee or is an employee of a third-party organizations involved in the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Rivera, CPI, Principal Investigator — Study PI
Locations (2):
- United States (2):
  - South Fla. Family Health & Research Ctr.LLC, Miami, Florida
  - Lice Source Services, Inc., Plantation, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eertmans F, Rossel B, Serrano L, Rivera E, Adriaens E. Efficacy and Safety of a Water-Based Head Lice Lotion: A Randomized, Controlled, Investigator-Blinded, Comparative, Bicentric Study. Dermatol Ther (Heidelb). 2019 Mar;9(1):143-157. doi: 10.1007/s13555-018-0274-x. Epub 2018 Nov 30. PMID 30506361

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Product | Reference
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Test Product: Water-based lotion (medical device)
- Reference: RID Shampoo
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 29 | 56
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Years | 15.3 (12.3) | 13.1 (10.9) | 14.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 33 | 68
  Not Hispanic or Latino | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 35 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70
Patients with at least 5 head lice and 5 living nits [Count of Participants; unit: Participants] | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Are Lice-free After 2 Treatments With Test Product (Including All Baseline Infestations).
Description: Clinical efficacy is reflected by the % of subjects that are lice-free after 2 topical applications (at day 0 & day 7 respectively) of the test product. In this analysis, all baseline infestations (mild, moderate, severe) have been included. Assessment is performed at study end (visit 4, day 10).
  A mild infestation corresponds to 5-9 lice and/or nymphs A moderate infestation corresponds to 10-24 lice and/or nymphs A severe infestation corresponds to 25 or more lice and/or nymphs
Time Frame: Day10
Population: In the first analysis, all subjects treated with the test product (n=35), have been analyzed (no correction for re-infestation). In a second analysis, a correction for re-infestation, defined as (1) no adult lice or third-stage nymphs present following the first treatment, and (2) no more than two adult lice or third-stage nymphs found on day 10, has been performed. Results are indicated in the table below.
Measure: Count of Participants; unit: Participants
Groups:
- Test Product: Water-based lotion (internal code (X92001666))
Arm/Group | Test Product
Number analyzed (Participants) | 35
Participants
  Number of lice-free subjects (uncorrected for re-infestation) | 30
  Number of lice-free subjects (corrected for re-infestation): number analyzed (Participants) | 34
  Number of lice-free subjects (corrected for re-infestation) | 30
Statistical Analysis 1: Comparison: Test Product; Efficacy analyses is performed on the ITT population (all subjects who were included and randomized in the study, with available baseline value of the primary endpoint and at least one follow-up visit). All statistical tests are performed at a 5% level of significance. The aim of this analysis is to show superiority for the cure rate of the test product versus a predefined limit of 70%. The following null hypothesis will be tested: H0, prim: pT - pR = 0 and Ha: pT - pR > 15% I; Test type: Superiority — In case superiority is not proven, non-inferiority is tested. As non-inferiority margin (δ), a 7.5% worse cure rate is regarded as clinically not relevant. The following null hypothesis will be used: H0, NI: pT-pR < δ, whereby δ = -7.5%. The lower, 95% confidence interval of the difference pT-pR will be used for the test. If H0, NI will be rejected, non-inferiority cannot be shown; p = 0.023, Chi-squared — A priori treshold p value of 0.05 for statistical significance was set prior to study start

2. Secondary Outcome: Number of Subjects That Are Lice-free After 2 Treatments With Reference Product (Including All Baseline Infestations).
Description: Clinical efficacy is reflected by the % of subjects that are lice-free after 2 topical applications (at day 0 & day 7 respectively) of the reference product. In this analysis, all baseline infestations (mild, moderate, severe) have been included. Assessment is performed at study end (visit 4, day 10).
  A mild infestation corresponds to 5-9 lice and/or nymphs A moderate infestation corresponds to 10-24 lice and/or nymphs A severe infestation corresponds to 25 or more lice and/or nymphs
Time Frame: Day 10
Population: In the first analysis, all subjects treated with the reference product (n=35), have been analyzed (no correction for re-infestation). In a second analysis, a correction for re-infestation, defined as (1) no adult lice or third-stage nymphs present following the first treatment, and (2) no more than two adult lice or third-stage nymphs found on day 10, has been performed. Results are indicated in the table below.
Measure: Count of Participants; unit: Participants
Groups:
- Reference Product: RID Shampoo (pyrethrum-based)
Arm/Group | Reference Product
Number analyzed (Participants) | 35
Participants
  Number of lice-free subjects (uncorrected for re-infestation) | 13
  Number of lice-free subjects (corrected for re-infestation): number analyzed (Participants) | 32
  Number of lice-free subjects (corrected for re-infestation) | 13

3. Secondary Outcome: Number of Subjects That Are Lice-free After 2 Treatments With Test Product (Only Mild and Moderate Baseline Infestations).
Description: The % of subjects with a mild (5-9 lice and/or nymphs) and moderate (10-24 lice and/or nymphs) baseline infestation that are lice-free after two topical treatments (day 0 & day 7) with the test product; assessed at study end (visit 4; day 10).
Time Frame: Day 10
Population: 28 subjects with light to moderate infestation (5-25 lice) and treated with test product have been included in this analysis. Subjects with severe infestation (>25 lice; n=7) were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product
Number analyzed (Participants) | 28
Participants | 25

4. Secondary Outcome: Number of Subjects That Are Lice-free After 2 Treatments With Reference Product (Only Mild and Moderate Baseline Infestations).
Description: The % of subjects with a mild (5-9 lice and/or nymphs) and moderate (10-24 lice and/or nymphs) baseline infestation that are lice-free after two topical treatments (day 0 & day 7) with the reference product; assessed at study end (visit 4; day 10).
Time Frame: Day 10
Population: 33 subjects with mild to moderate infestation, treated with reference product, have been included in this analysis. Subjects with severe infestation (>25 lice; n=2) were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference
Number analyzed (Participants) | 33
Participants | 13

5. Secondary Outcome: Number of Subjects That Are Lice-Free After 1 Treatment With Test Product (All Baseline Infestations).
Description: The % of subjects that are lice-free after one topical treatment with the test product (assessment 24h post treatment), considering all baseline infestations (mild, moderate, severe).
  A mild infestation corresponds to 5-9 lice and/or nymphs A moderate infestation corresponds to 10-24 lice and/or nymphs A severe infestation corresponds to 25 or more lice and/or nymphs
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product
Number analyzed (Participants) | 35
Participants | 30

6. Secondary Outcome: Number of Subjects That Are Lice-free After 1 Treatment With Reference Product (All Baseline Infestations).
Description: The % of subjects that are lice-free after one topical treatment with the reference product (assessment 24h post treatment), considering all baseline infestations (mild, moderate, severe).
  A mild infestation corresponds to 5-9 lice and/or nymphs A moderate infestation corresponds to 10-24 lice and/or nymphs A severe infestation corresponds to 25 or more lice and/or nymphs
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Reference
Number analyzed (Participants) | 35
Participants | 21

7. Secondary Outcome: Effect of Both Investigational Treatments on Pruritus (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator.
Description: The occurrence and degree of pruritus is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: the scalp does not itch; Mild: occasional episodes of itching, not bothersome; Moderate: frequent, several times a day, bothersome; Severe: nearly constant, frequent scratching, very bothersome.
Time Frame: Day 0, Day 1, Day 7, Day10
Population: Concerns a safety parameter. The safety set/population consists of all subjects who were randomised and exposed to study medication. The table below shows the total number of participants in each test group, experiencing mild to severe pruritus (combined), at the different evaluation time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference
Number analyzed (Participants) | 35 | 35
Participants
  Pruritus D0 pre-treatment | 27 | 24
  Pruritus D0 post-treatment | 14 | 13
  Pruritus D1 | 8 | 5
  Pruritus D7 pre-treatment | 9 | 8
  Pruritus D7 post-treatment | 4 | 3
  Pruritus D10 | 7 | 5

8. Secondary Outcome: Effect of Both Investigational Treatments on Scalp Excoriation (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator.
Description: The occurrence and degree of scalp excoriation (breaking of the skin, usually caused by scratching) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no broken skin on the scalp; Mild: one or two areas on the scalp on which skin is broken; Moderate: more than two separate areas of the scalp with broken skin but not generalized across the scalp; Severe: widespread breaking of the skin involving most of the scalp.
Time Frame: Day 0, Day 1, Day 7, Day10
Population: Concerns a safety parameter. The safety set/population consists of all subjects who were randomised and exposed to study medication. The table below shows the total number of participants in each test group, experiencing mild to severe scalp excoriation (combined), at the different evaluation time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference
Number analyzed (Participants) | 35 | 35
Participants
  Scalp Excoriation D0 pre-treatment | 0 | 0
  Scalp Excoriation D0 post-treatment | 0 | 0
  Scalp Excoriation D1 | 0 | 0
  Scalp Excoriation D7 pre-treatment | 0 | 0
  Scalp Excoriation D7 post-treatment | 0 | 0
  Scalp Excoriation D10 | 0 | 0

9. Secondary Outcome: Effect of Both Investigational Treatments on Paraesthesia (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator.
Description: The occurrence and degree of paraesthesia (tingling or prickling sensation) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no tingling or prickling sensation; Mild: occasional tingling or prickling sensation; Moderate: frequent tingling or prickling sensation; Severe: nearly constant tingling or prickling sensation
Time Frame: Day 0, Day 1, Day 7, Day10
Population: Concerns a safety parameter. The safety set/population consists of all subjects who were randomised and exposed to study medication. The table below shows the total number of participants in each test group, experiencing mild to severe paraesthesia (combined), at the different evaluation time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference
Number analyzed (Participants) | 35 | 35
Participants
  Paraesthesia D0 pre-treatment | 0 | 0
  Paraesthesia D0 post-treatment | 0 | 0
  Paraesthesia D1 | 0 | 0
  Paraesthesia D7 pre-treatment | 0 | 0
  Paraesthesia D7 post-treatment | 0 | 0
  Paraesthesia D10 | 0 | 0

10. Secondary Outcome: Effect of Both Investigational Treatments on Skin Erythema (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator.
Description: The occurrence and degree of skin erythema (redness of the scalp) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no redness of the scalp; Mild: faint, barely perceptible erythema with limited distribution; Moderate: diffuse pink areas of scalp are readily visible; Severe: large areas of the scalp are red.
Time Frame: Day 0, Day 1, Day 7, Day10
Population: Concerns a safety parameter. The safety set/population consists of all subjects who were randomised and exposed to study medication. The table below shows the total number of participants in each test group, experiencing mild to severe skin erythema (combined), at the different evaluation time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference
Number analyzed (Participants) | 35 | 35
Participants
  Skin erythema D0 pre-treatment | 0 | 1
  Skin erythema D0 post-treatment | 0 | 1
  Skin erythema D1 | 0 | 1
  Skin erythema D7 pre-treatment | 0 | 0
  Skin erythema D7 post-treatment | 0 | 0
  Skin erythema D10 | 0 | 0

11. Secondary Outcome: Effect of Both Investigational Treatments on Pyroderma (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator.
Description: The occurrence and degree of pyroderma (sores filled with clear fluid, pus or crusting) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no lesions visible on the scalp; Mild: one or two lesions visible with crusting or other evidence of infection; Moderate: presence of more than two lesions with crusting or other evidence of infection, but not generalized across the scalp; Severe: lesions with crusting or other evidence of infection, involving most of the scalp.
Time Frame: Day 0, Day 1, Day 7, Day10
Population: Concerns a safety parameter. The safety set/population consists of all subjects who were randomised and exposed to study medication. The table below shows the total number of participants in each test group, experiencing mild to severe pyroderma (combined), at the different evaluation time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference
Number analyzed (Participants) | 35 | 35
Participants
  Pyroderma D0 pre-treatment | 0 | 1
  Pyroderma D0 post-treatment | 0 | 0
  Pyroderma D1 | 0 | 0
  Pyroderma D7 pre-treatment | 0 | 0
  Pyroderma D7 post-treatment | 0 | 0
  Pyroderma D10 | 0 | 0

12. Secondary Outcome: Effect of Both Investigational Treatments on Eye Irritation, as Assessed by a Blinded Clinical Investigator.
Description: The occurrence and degree of eye irritation (stinging, burning sensation, and/or pain) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no stinging, burning or pain Mild: slight mild stinging, burning or pain Moderate: moderate stinging, burning or pain Severe: severe stinging, burning or pain
Time Frame: Day 0, Day 1, Day 7, Day10
Population: Concerns a safety parameter. The safety set/population consists of all subjects who were randomised and exposed to study medication. The table below shows the total number of participants in each test group, experiencing mild to severe eye irritation (combined), at the different evaluation time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference
Number analyzed (Participants) | 35 | 35
Participants
  Eye irritation D0 pre-treatment | 0 | 0
  Eye irritation D0 post-treatment | 0 | 0
  Eye irritation D1 | 0 | 0
  Eye irritation D7 pre-treatment | 0 | 0
  Eye irritation D7 post-treatment | 0 | 0
  Eye irritation D10 | 0 | 0

13. Secondary Outcome: Global Tolerability, Evaluated at Study End (Visit 4, Day 10)
Description: Global tolerability is defined as the general well-being and comfort of the subjects. This parameter is assessed at day 10 in subjects, treated with either test product or reference product, respectively. The subject is asked to score his general feeling at study end and must provide a justification for his/her answer. Scoring was performed as follows: very good (best case), good, moderate, or poor (worst case).
Time Frame: Day 10
Population: All subjects that have been treated at D0 & D7 with test or reference product, respectively.
Measure: Count of Participants; unit: Participants
Groups:
- Test Product: Evaluation of erythema, paraesthesia, excoriations, pyrodema, puritus and abnormalities
Arm/Group | Test Product | Reference
Number analyzed (Participants) | 35 | 35
Participants
  Very good | 23 | 17
  Good | 12 | 18

14. Other Pre Specified Outcome: Assessment of Adverse Events Occurring After 1 and 2 Treatments With Both Investigational Products.
Description: Recording Adverse Events and investigating the relationship with the treatment. At each visit (D0: first treatment; D1: 24h post-treatment assessment; D7: second treatment; D10: final assessment), the clinical staff is recording adverse events (if any) and evaluates the correlation with the treatment.
Time Frame: Study period (10 days) + in case of adverse events: clinical staff will monitor the trial subject's safety from the occurrence of an AE until recovery, return to baseline or a stable state will be achieved.
Population: All subjects that have been exposed to at least 1 treatment (either test product or reference).
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference
Number analyzed (Participants) | 35 | 35
Participants
  All-cause mortality | 0 | 0
  Serious Adverse Events | 0 | 0
  Other Adverse Events (Not including serious AE) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are recorded over the period of the clinical trial (10 days per subject). Furthermore, the study staff must monitor the trial subject's safety from the occurrence of an AE until recovery, return to baseline or a stable state will be achieved. In single cases, follow up of an AE/SAE after last visit can be omitted if there is no causal relationship to study drug and subject's state is improved or stabilized.
Description: No difference in definition
Arm/Group | Test Product | Reference
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

LIMITATIONS AND CAVEATS:
Limitations of this study:

1. Moderate number of subjects.
2. Reference product: instead of a pyrethroid-based product, a silicone-based pediculicide might have served as reference.
3. No subgroup analyses performed to evaluate the impact of infestation degree, hair characteristics, & other parameters. However, no remarkable differences found in baseline parameters between both groups.
4. Dry combing to diagnose a head lice infestation (may be less sensitive compared to wet combing).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT03617926/Prot_SAP_000.pdf